CLINICAL TRIAL: NCT04835558
Title: Respiratory Muscle Endurance in Obesity Hypoventilation Syndrome; Evaluation by Incremental Load Test
Brief Title: Respiratory Muscle Endurance in Obesity Hypoventilation Syndrome
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Goksen Kuran Aslan, Assoc. Prof., Istanbul University - Cerrahpasa
Other Study IDs: 29713
Record Dates: First submitted 2021-03-28; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Obesity Hypoventilation Syndrome (OHS)
Keywords: Respiratory Muscle Endurance; Sleep; Fatigue; Quality of Life
MeSH Terms: conditions — Obesity Hypoventilation Syndrome; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: Subjects with obesity hypoventilation sydrome (30 < body mass index < 40 kg/m2)
- Group II: Subjects with obesity hypoventilation sydrome (body mass index > 40 kg/m2)
- Control Group: Age and sex-matched obese subjects (30 < body mass index < 40 kg/m2) with low risk of obstructive sleep apnea (STOP-BANG score < 3)

SUMMARY:
Obesity hypoventilation syndrome (OHS) is defined as a combination of obesity [body mass index (BMI) ≥30 kg/m2], chronic daytime hypercapnia (PaCO2 >45 mm Hg), and sleep-apnea in the absence of other known causes of hypercapnia. Respiratory system compliance decreases and resistance increases in OHS. This causes increase in work of breathing and oxygen cost of breathing, which may result in respiratory muscle fatigue. Increase in respiratory workload and increase in resistance to respiration is expected to decrease in respiratory muscle endurance (RME) in subjects with OHS.

DETAILED DESCRIPTION:
In the literature, studies evaluating RME in subjects with OHS are limited. No study has been found to evaluate RME using the incremental load test in subjects with OHS. Accordingly, it was aimed to evaluate and compare respiratory muscle endurance in subjects with OHS and a control group, and to determine factors associated with respiratory muscle endurance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with OHS
* Obese subjects (30 < body mass index < 40 kg/m2) with low risk of obstructive sleep apnea (STOP-BANG score < 3)

Exclusion Criteria:

* Severe respiratory disease
* Subjects with orthopeadic and/or neurologic disorders that could limit exercise tests

Ages: 24 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who had polysomnography performed in the sleep laboratory and were diagnosed with OHS were screened.
  Age and sex-matched obese subjects (30 < body mass index < 40 kg/m2) with low risk of obstructive sleep apnea (STOP-BANG score < 3) included in the study as the control group.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Incremental load test | 1 day
  Respiratory muscle endurance was evaluated by incremental load test. The incremental load test was performed using the electronic inspiratory loading device (PowerBreathe®-KHP2).

SECONDARY OUTCOMES:
Mouth pressure measurements | 1 day
  Respiratory muscle strength was measured using mouth pressure measurements (Micro Medical MicroRPM).
6 minute walk test | 1 day
  The 6 minute walk test was used to evaluate the functional exercise capacity of the subjects.
Epworth Sleepiness Scale | 1 day
  Excessive daytime sleepiness was assessed with the Epworth Sleepiness Scale. A score of >10 accepted as daytime sleepiness.
Pittsburg Sleep Quality Index | 1 day
  Sleep quality was assessed with the Pittsburg Sleep Quality Index. The total score were interpreted as follows: 0-5 indicated good sleep quality, > 5 indicated poor sleep quality, and >10 indicated the presence of a sleep disorder.
Fatigue Severity Scale | 1 day
  Fatigue severity was assessed with the Fatigue Severity Scale. This seven-likert scale was used for each item and final score was accepted as mean value of the 9 items. The higher scores indicated higher fatigue severity.
EQ-5D Health-Related Quality of Life Questionnaire | 1 day
  Quality of life was assessed with the EQ-5D Health-Related Quality of Life Questionnaire. The maximum score of 1 indicates the best health state, and higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status in which 100 indicates the best health status.
Obesity and Weight Loss Quality of Life Instrument | 1 day
  Quality of life specific to obesity was assessed with the Obesity and Weight Loss Quality of Life Instrument. As the total score from the scale approaches 0, the quality of life decreases, and as it approaches 100, the quality of life increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)